CLINICAL TRIAL: NCT01017575
Title: A Phase 2a Study of Daclatasvir in Combination With Peginterferon Alfa-2a(Pegasys®) and Ribavirin (Copegus®) in Japanese Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Safety and Efficacy of Daclatasvir (BMS-790052) Plus Standard of Care in Japanese Patients (Pegylated-interferon Alpha-2a and Ribavirin)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI444-022
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin) (Experimental): Treatment Naive
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm B (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin) (Experimental): Treatment Naive
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm C (Placebo, plus Peginterferon alfa-2a, Ribavirin) (Placebo Comparator): Treatment Naive
  Interventions: Drug: Placebo; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm D (Daclatasvir, plus peginterferon alfa-2a, Ribavirin) (Experimental): Non-Responder
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Arm E (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin) (Experimental): Non-Responder
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Tablets, Oral, 10 mg, daily, 24-48 weeks
  Arms: Arm A (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin); Arm D (Daclatasvir, plus peginterferon alfa-2a, Ribavirin)
Drug: Daclatasvir — Tablets, Oral, 60 mg, daily, 24-48 weeks
  Arms: Arm B (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin); Arm E (Daclatasvir, plus Peginterferon alfa-2a, Ribavirin)
Drug: Placebo — Tablets, Oral, 0 mg, daily, 48 weeks
  Arms: Arm C (Placebo, plus Peginterferon alfa-2a, Ribavirin)
Drug: Peginterferon alfa-2a — Syringe, Subcutaneous, 180µg, weekly, 24-48 weeks
  Other Names: Pegasys®
Drug: Ribavirin — Tablets, Oral, 600 to 1000 mg based on weight, daily, 24-48 weeks
  Other Names: Copegus®

SUMMARY:
The purpose of this study is to identify at least 1 dose of Daclatasvir, that when combined with peginterferon-alfa (PegIFNα) and ribavirin (RBV) for the treatment of chronically infected HCV genotype 1 treatment-naïve and non-responder to standard of care subjects is safe, well tolerated, and efficacious

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects chronically infected with hepatitis C virus (HCV) genotype 1
* HCV RNA viral load ≥ 10*5* IU/mL (100,000 IU/mL) at screening
* The current standard of care naïve or non-responder

Key Exclusion Criteria:

* Cirrhosis
* HCC
* Co-infection with hepatitis B virus (HBV), HIV-1 or HIV-2

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Japan (5):
  - Local Institution, Chiba, Chiba
  - Local Institution, Kurume-Shi, Fukuoka
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Musashino-Shi, Tokyo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in Japan.
Pre-assignment Details: A total of 55 participants were enrolled, of which 43 participants were randomized and 42 were treated. 12 participants were not randomized because 10 no longer met study criteria and 2 withdrew consent; 1 randomized participant was not treated due enlarged lymph node.
Groups:
- Placebo+pegIFNα-2a+Ribavirin (Treatment Naive): Participants received a matching placebo of daclatasvir tablet, orally, once daily (OD) with peginterferon alpha-2a (pegIFNα-2a) subcutaneously once weekly and ribavirin orally, twice daily (BID). Treatment naive participants were those who had never been exposed to any Hepatitis C Virus (HCV) therapy with interferon (IFN) -containing regimens including pegIFNα-2a/ ribavirin.
- Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive): Participants received 10-mg of daclatasvir OD coadministered with pegIFNα-2a subcutaneously once weekly and ribavirin orally BID. Treatment naive participants were defined as those who had never been exposed to any HCV therapy with IFN- containing regimens including pegIFNα-2a/ ribavirin.
- Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive): Participants received 60-mg of daclatasvir OD coadministered with pegIFNα-2a administered subcutaneously once weekly and ribavirin administered orally BID. Treatment naive participants were defined as those who had never been exposed to any HCV therapy with IFN- containing regimens including pegIFNα-2a/ ribavirin.
- Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders): Participants received 10-mg of daclatasvir OD coadministered with pegIFNα-2a subcutaneously once weekly and ribavirin orally BID. Non-responders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα-2a/ ribavirin.
- Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders): Participants received 60-mg of daclatasvir OD coadministered with pegIFNα-2a administered subcutaneously once weekly and ribavirin administered orally BID. Non-responders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα-2a/ ribavirin.
Period: Overall Study
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Started | 8 | 9 | 8 | 8 | 9
Completed | 7 | 7 | 8 | 7 | 6
Not Completed | 1 | 2 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants who received at least 1 dose of study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Total
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 42
Age, Customized [Number; unit: participants]
  <65 years | 7 | 8 | 6 | 6 | 8 | 35
  >=65 years | 1 | 1 | 2 | 2 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 2 | 4 | 22
  Male | 3 | 4 | 2 | 6 | 5 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as undetectable hepatitis C virus (HCV) RNA ie, HCV RNA <15 IU/mL, the lower limit of detection at Week 4.
Time Frame: Week 4
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
percentage of participants | 12.5 | 77.8 | 62.5 | 62.5 | 88.9

2. Secondary Outcome: Percentage of Participants With a Complete Early Virologic Response (cEVR)
Description: cEVR was defined as hepatitis C virus RNA <15 IU/mL at Week 12.
Time Frame: Week 12
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
percentage of participants | 62.5 | 88.9 | 100 | 87.5 | 88.9

3. Secondary Outcome: Percentage of Participants With a Sustained Virologic Response (SVR) at Follow-up Week 12 and Follow-up Week 24
Description: SVR at Follow-up Week 12 (SVR12) and SVR at Follow-up week 24 (SVR24) was defined as hepatitis C virus (HCV) RNA <15 IU/mL at follow-up Weeks 12 and 24.
Time Frame: Follow up Week 12, Follow up Week 24
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
percentage of participants
  SVR12 | 75 | 88.9 | 100 | 50 | 77.8
  SVR24 | 75 | 88.9 | 100 | 50 | 77.8

4. Primary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as undetectable hepatitis C virus (HCV) RNA ie, HCV RNA <15 IU/mL, the lower limit of detection at both Weeks 4 and 12.
Time Frame: From Week 4 up to Week 12
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
percentage of participants | 12.5 | 66.7 | 62.5 | 62.5 | 77.8

5. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), and Who Died.
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not has a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From Baseline up to 30 days after last dose of study drug
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
participants
  SAEs | 0 | 2 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 1 | 0 | 0 | 2
  Death | 0 | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities
Description: Clinically significant change in marked laboratory abnormalities (Grade 3 to 4) included: Aspartate aminotransferase (AST)- Grade 3 as >5.0 to 10.0*Upper Limit of Normal (ULN), Grade 4 as >10.0*ULN; Hemoglobin- Grade 3 as 7.0 to 8.9 g/dL, Grade 4 as <7.0 g/dL; Neutrophils- Grade 3 as 0.5 to 0.749*10^9/L, Grade 4 as <0.5*10^9/L; Lymphocytes- Grade 3 as 0.35 to 0.499*10^9/L, Grade 4 as <0.35*10^9/L; Platelets- Grade 3 as 25000 to 49999*10^9/L, Grade 4 as <25000 10^9/L; white blood cells (WBC) - Grade 3 as 1000 to 1499*10^9/L, Grade 4 as <1000*10^9/L and Lipase- Grade 3 as 3.1-5.0*ULN, Grade 4 as >5.0*ULN.
Time Frame: From screening up to Week 12 (treatment period)
Population: All treated participants who received at least 1 dose of study therapy.
Measure: Number; unit: Participants
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9
Participants
  Hemoglobin | 0 | 2 | 1 | 0 | 2
  Lymphocytes | 5 | 2 | 4 | 5 | 3
  Neutrophils | 4 | 4 | 3 | 3 | 2
  Platelets | 0 | 0 | 0 | 2 | 0
  WBC | 3 | 1 | 2 | 2 | 2
  AST | 0 | 0 | 0 | 1 | 0
  Lipase | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders)
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/9 | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8 | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) (N=9) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) (N=8) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders) (N=9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+pegIFNα-2a+Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Treatment Naive) (N=9) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin (Non-Responders) (N=8) | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin (Non-Responders) (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 3
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 3 | 2 | 3
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Retinopathy (Eye disorders) | 1 | 2 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 3 | 5 | 2 | 3
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 5 | 4 | 5
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 5 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 4 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Body temperature decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Eyelids pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 4 | 2 | 3 | 2
Feeling abnormal (General disorders) | 0 | 1 | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 1
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 5 | 6 | 5 | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 2 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 2 | 3
Chills (General disorders) | 4 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2 | 4 | 5 | 3
Malaise (General disorders) | 5 | 1 | 4 | 2 | 5
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 3 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 4
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 5
Dysgeusia (Nervous system disorders) | 1 | 2 | 2 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 3 | 3 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Administration site reaction (General disorders) | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 0 | 4 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 1 | 2 | 0 | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 2
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Retinal exudates (Eye disorders) | 2 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single center publications until after disclosure of the clinical trial's primary publication.